CLINICAL TRIAL: NCT01361165
Title: Data Analysis for 04-C-0234 Tenofovir Disoproxil Fumarate Salvage Therapy in HIV-Infected Children and a Study of Its Effect on Bone Metabolism
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999906255; 06-C-N255
Record Dates: First submitted 2011-05-24; First posted 2011-05-26 (Estimated); Last update posted 2023-10-31 (Actual); Status verified 2011-05

CONDITIONS: HIV-Infected Children
Keywords: Pediatric; Data Analysis

SUMMARY:
We plan to analyze the data to meet the primary objective of the study:

To characterize the change in bone mineral density (BMD), as measured by lumbar spine DEXA, during and following treatment with tenofovir DF-containing antiretroviral therapy in HIV-infected children.

In addition, we plan to analyze the data to meet 2 secondary objectives of the study:

1. To study and monitor markers of bone metabolism - calcium, phosphorus, parathyroid hormone (PTH), vitamin D levels, bone resorption markers (urinary collagen cross-linked N-telopeptide and free deoxypyridinoline), bone formation markers (bone specific alkaline phosphatase and osteocalcin) - in HIV-infected children treated with tenofovir DF-containing antiretroviral therapy.
2. To study immunologic, virologic and clinical effects of tenofovir DF administered to HIV-infected children in combination with other antiretroviral therapies.

DETAILED DESCRIPTION:
We plan to analyze the data to meet the primary objective of the study:

To characterize the change in bone mineral density (BMD), as measured by lumbar spine DEXA, during and following treatment with tenofovir DF-containing antiretroviral therapy in HIV-infected children.

In addition, we plan to analyze the data to meet 2 secondary objectives of the study:

1. To study and monitor markers of bone metabolism - calcium, phosphorus, parathyroid hormone (PTH), vitamin D levels, bone resorption markers (urinary collagen cross-linked N-telopeptide and free deoxypyridinoline), bone formation markers (bone specific alkaline phosphatase and osteocalcin) - in HIV-infected children treated with tenofovir DF-containing antiretroviral therapy.
2. To study immunologic, virologic and clinical effects of tenofovir DF administered to HIV-infected children in combination with other antiretroviral therapies.

ELIGIBILITY:
* Data Analysis Only

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2006-09; Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States